CLINICAL TRIAL: NCT02579109
Title: Exploring Social Cognition in Autism Spectrum Disorder With Long Time Memory Task. Controlled Study on 8-13 Years Childs
Brief Title: Multisensorial Information's Treatment in Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13AOI09
Record Dates: First submitted 2015-09-29; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- autistic patient (Other): patient with autistic trouble
  Interventions: Other: memory test
- healthy volunteers (Other): healthy volunteers
  Interventions: Other: memory test

INTERVENTIONS:
Other: memory test

SUMMARY:
Introduction:

Autism spectrum disorder is characterized by deficits in three functional domains: language and communication, social reciprocity, and the presence of restricted interests/repetitive behaviors. There's also deficits in social cognition. When having a face-to-face conversation, a listener not only hears what a speaker is saying, but also sees the articulatory gestures that accompany those sounds. Speech signals needs then a multisensory processing. Impairments in multisensory perceptual binding may be particularly relevant in ASD, given that hallmark features of the disorder include difficulties in speech, communication, and social interactions.

Objectives:

The investigator suggest that atypical multisensory processing in ASD may have an impact on speech perception and social processing.

Aims:

Methods:

This pilot study measures free recall scores in 3 lists of words presentation after 30 minutes. In the first condition (CI) words are only listening. In the second condition (CII) words are associated with a picture of a mans face. In the third condition (CIII) words are associated with a video of a man speaking. Three lists are homogeneous form words characteristics (lexical frequency, emotional valence norm, imageability). Participants were 7- to 13-year-olds typically developing children (TD) (N = 19) and ASD children (N = 19).

The investigator would create some new tools for exploring the treatment of a social information. These tools should be the closest of a ecological social interaction.

ELIGIBILITY:
Inclusion Criteria:

* Boy or girl,
* 7 - 13 years,
* Presenting a diagnosis DSM IV of disorder(confusion) of the autistic spectre: detected by the scale(ladder) ADI ( Autism Diagnostic Interview) or by TEENAGERS (Autism Diagnostic Observation Schedule): typical autistic. These patients do not answer the diagnosis of psychosis according to Kiddie-SADS,
* Upper total IQ or equal to 50, examination dating less than year before the inclusion,
* French-speaking children,
* Signature of the informed consent by the parents(relatives) and the child,
* Membership to the Social Security.

Exclusion Criteria:

* Genetic, neurological or neurosensory pathologies,
* Diagnosis of intrusive disorder(confusion) of the not specified development: TED our,
* The patients will not be included who would participate in a program or a study of reeducation in the social fitnesses.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
rate of reminder after 30 minutes between the group autistic and the group witness( %) | 30 minutes
  Comparison between the group autistic and the group witness of the difference enter the rate of reminder(abseiling) in 30 minutes of the words proposed in video and audio sequences.

SECONDARY OUTCOMES:
Difference of the scores of reminders words (%) | 30 minutes
  Difference of the scores of reminders between the both group, immediately after procedure and 30 minutes after procedure